CLINICAL TRIAL: NCT00681278
Title: A Retrospective, Multi Centre, Non-interventional, Observational Study to Investigate Treatment Pattern of Blood Pressure in the Type II Diabetes Mellitus Patients With Hypertension.
Brief Title: Retrospective Survey for Patients With Hypertension and Diabetes Mellitus
Acronym: CRYSTAL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Joon Woo Bahn, AstraZeneca
Other Study IDs: NIS-CKR-DUM-2008/2
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-12

CONDITIONS: Hypertension
Keywords: Hypertension; Type II DM; JNC7; 2007 ESH-ESC guidelines; survey
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- 1: Hypertension patients with Type II Diabetes mellitus

SUMMARY:
This study will address the treatment rate and control rate of hypertension, treatment pattern and factors to affect blood pressure control by examining (retrospective) medical records of hypertension patients having Type 2 Diabetes mellitus, among outpatients coming to the Endocrinology Department in 20 general hospital settings nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient Type II DM patients receiving hypertension medication in 2006
* Patient with Type II DM receiving hypertension medication during at least 1 year.

Exclusion Criteria:

* Secondary hypertension patients
* Patients not receiving hypertension medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with type II Diabetes mellitus, receiving hypertension medication during at least 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Attainment rate to the target blood pressure. | After collecting all Patient Record Form.

SECONDARY OUTCOMES:
Dropout rate will be estimated during the follow-up period after the hypertension treatment. Attainment to the target blood pressure will be investigated according to concomitant diseases. | After collecting all Patient Record Form.
Change in DBP/SBP value during the follow-up period will be addressed. Change in the DBP/SBP value will be investigated according to the risk factors and concurrent disease. | After collecting all Patient Record Form.

CONTACTS AND LOCATIONS:
Overall Officials: Joon Woo Bahn, Study Director — Astrazenca Korea medical dept,.
Locations (13):
- South Korea (13):
  - Research Site, Bucheon-si, Gyeonggi-do
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Guri-si, Gyeonggi-do
  - Research Site, Sungnam, Gyeonggi-do
  - Research Site, Jeonju, Keollabuk
  - Research Site, Busan
  - Research Site, Deagu
  - Research Site, Deajeon
  - Research Site, Incheon
  - Research Site, Kwangju
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Wŏnju